CLINICAL TRIAL: NCT01603680
Title: Circumferential Versus Not Circumferential Distribution of Mepivacaine Around the Median and Ulnar Nerves in the Carpal Tunnel Surgery. Randomized Clinical Trial, Double Blinded.
Brief Title: Distribution Circumferential Versus Non Circumferential of Mepivacaine in the Median and Ulnar Nerves
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Principal Investigator, Paula Diéguez García, Principal Investigator, Complexo Hospitalario Universitario de A Coruña
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ArAL 11.1; 2011-002608-34 (EudraCT Number)
Record Dates: First submitted 2012-01-16; First posted 2012-05-22 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Anesthesia
Keywords: Ultrasonography; Block nerve; Anaesthesia; Carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Circumferential (C) (Other): "Circumferential"(C) spread group will be defined as mepivacaine injectate visualized by ultrasonography all around the median and ulnar nerves imaged in short axis.
  Interventions: Procedure: Circumferential spread of the mepivacaine ultrasonographic guided around the median and ulnar nerves at the elbow
- Non circumferential (NC) (Other): Local anesthetic spread will be asymmetrical around the median and ulnar nerves, the mepivacaine will be partially in contact with the nerve
  Interventions: Procedure: Non circumferential spread in ultrasound-guided median and ulnar nerves block

INTERVENTIONS:
Procedure: Circumferential spread of the mepivacaine ultrasonographic guided around the median and ulnar nerves at the elbow — Homogeneous spread of 6 ml of mepivacaine 1% around the median and ulnar nerves in each one using several needle passes and active hydrodissection
  Other Names: Local anesthetic spread; "Doughnut sign"
  Arms: Circumferential (C)
Procedure: Non circumferential spread in ultrasound-guided median and ulnar nerves block — Asymmetric spread of 6 ml of mepivacaine 1% in contact with median and ulnar nerves block in each one, using only one needle pass
  Other Names: Asymmetric local anesthetic spread
  Arms: Non circumferential (NC)

SUMMARY:
1. Evaluation of the efficacy of the circumferential versus non circumferential distribution of mepivacaine around the median and ulnar nerves.
2. Evaluation the onset of action of mepivacaine in circumferential versus non circumferential distribution around the median and ulnar nerves.
3. Spread of mepivacaine after injection guided by ultrasonography.
4. Complications of both anesthetic techniques in postoperative time.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled patients for surgery of carpal tunnel including patients in ASA I-III status, without exclusion criteria. The principal investigator study and/or other designated site staff will obtain written informed consent from all research patients.

Exclusion Criteria:

* Abnormal bleeding, infection in the punction side, allergy or other problems with the medication of the study, muscular or nerve diseases, patients < 18 years old, pregnancy, cognitive disease or reject of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Efficacy and onset of action | On arrival in the recovery room
  Sensory block will be assessed as a loss of cold sensation elicited by a cold wet cotton swab in the areas of the medial and ulnar nerves by comparison with contralateral hand. Sensory block will be clasiffied as follows: 0, anesthesia; 1, hyposthesia; 2, normal sensation. Motor function will be tested as according to a modified Bromage score: 0, no motor blokade; 1, weak response against resistence; 2, complete motor blockade. Motor and sensory blockades will be assessed by a blinded observer at 5, 15, 30 mins after local anesthetic injection and on arrival in the recovery room.

SECONDARY OUTCOMES:
Complications in postoperative time | 24 hours postoperative time
  Since the nerve block to the hospital outcome will be registered potencial block-related complications. At the first postoperative day, each patient will be called by phone, to report the time at first onset of pain in the operative site and lack of residual postoperative neurologic symptoms, postoperative nausea and vomiting, and hospital readmission (for severity of pain or bleeding or other reasons)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Diéguez, Anesthetist, Principal Investigator — Complexo Hospitalario Universitario A Coruña
Locations (1):
- Complexo Hospitalario Universitario A Coruña. Hospital Abente y Lago, A Coruña, A Coruña, Spain

REFERENCES:
- [Result] Al-Nasser B, Hubert C, Negre M. Role of local anesthetic spread pattern and electrical stimulation in ultrasound-guided musculocutaneous nerve block. J Clin Anesth. 2010 Aug;22(5):334-9. doi: 10.1016/j.jclinane.2009.09.008. PMID 20650379
- [Result] Morau D, Levy F, Bringuier S, Biboulet P, Choquet O, Kassim M, Bernard N, Capdevila X. Ultrasound-guided evaluation of the local anesthetic spread parameters required for a rapid surgical popliteal sciatic nerve block. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):559-64. doi: 10.1097/AAP.0b013e3181fa6b60. PMID 20975475
- [Derived] Dieguez-Garcia P, Lopez-Alvarez S, Juncal J, Lopez AM, Sala-Blanch X. Comparison of the effectiveness of circumferential versus non-circumferential spread in median and ulnar nerve blocks. A double-blind randomized clinical trial. Reg Anesth Pain Med. 2020 May;45(5):362-366. doi: 10.1136/rapm-2019-101157. Epub 2020 Mar 11. PMID 32165554